CLINICAL TRIAL: NCT01589575
Title: Evaluation of the Impact of Symptoms of Anxiety and Depression in Relatives of Critically Ill Patients: Spouses Versus Other Close Relatives
Brief Title: Anxiety and Depression in Relatives of Critically Ill Patients: Spouses Versus Other Close Relatives
Acronym: StressRéa
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2012/CR-03; 2012-A00501-42 (Other: RCB number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety; Depression
Keywords: Intensive Care Unit
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spouses: This group of relatives includes the spouses of ICU patients (over 16 years of age and intubated and under ventilation for at least 48 hours) meeting stated inclusion criteria.
- Other relatives: This group of relatives includes the non-spouse relatives of ICU patients (over 16 years of age and intubated and under ventilation for at least 48 hours) meeting stated inclusion criteria.

SUMMARY:
The main objective of this study is to compare the rate of reported anxiety / depression (HADS >= 8) among spouses and other family members in ICU patients.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* to assess symptoms of anxiety (HADS ≥ 8) and depression (HADS ≥ 8) among relatives of ICU patients three months after discharge
* to assess what relatives felt vis-à-vis the information process
* describe the number and duration of interviews with participants
* to compare variables between the groups "spouses" and "other relatives".

  * satisfaction
  * number and duration of interviews
  * HADS questionnaire
  * The scale Edmunton
  * an internal questionnaire
  * IES-R score
  * level of mental well-being: WEMWBS
* to describe the completeness of the study
* to test the hypothesis that the development of symptoms related to physical manifestations of anxiety and depression predicts the development of post-traumatic stress at 3 months.
* to assess the impact of the various forms of stress during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* The relative must have given his/her informed and signed consent
* The relative must be insured or beneficiary of a health insurance plan
* The relative must be available for 3 months of follow-up

Exclusion Criteria:

* The relative is under judicial protection, under tutorship or curatorship
* The relative refuses to sign the consent
* It is impossible to correctly inform the relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes relatives of patients admitted to intensive care (over the age of 16 years and intubated and ventilated for at least 48 hours). The study population mainly inclused spouses, parents, children, and siblings of patients in intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Presence/absence of a score >= 8 on the Hospital Anxiety and Depression Scale Questionnaire | 3 months after the patients is discharged from the ICU unit

SECONDARY OUTCOMES:
* Presence/absence of a score >= 8 on the Hospital Anxiety and Depression Scale Questionnaire | 4-6 days after the admission of a patient to the ICU
VAS score for satisfaction concerning the communication of information concerning the patient currently in the ICU | During the ICU stay (days 1 to 28)
  Visual Analog Scale ranging from 1 to 10
Number of interviews | During the ICU stay (days 1 to 28)
  Number of interviews the relative has with medical staff
Mean interview duration (minutes) | During the ICU stay (days 1 to 28)
Edmonton Symptom Assessment Scale Score | 4-6 days after the admission of a patient to the ICU
The Impact of Event Scale - Revised (IES-R) | 3 months after the patients is discharged from the ICU unit
The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | 3 months after the patients is discharged from the ICU unit

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France